CLINICAL TRIAL: NCT03925454
Title: FREquent DIalysis and Markers of Cardiac Strain and Injury, Physical Fitness, Habitual Physical Activity and Quality of Life: an Observational Pilot Study
Brief Title: FREquent DIalysis & Markers of Cardiac Strain and Injury, Physical Fitness, Habitual Physical Activity & Quality of Life
Acronym: FREDI-CAL
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: NxStage Medical (Other); University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2017/122
Record Dates: First submitted 2019-03-29; First posted 2019-04-24 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-Centre Haemodiafiltration (ICHDF) Group: Participants undergoing ICHDF treatment will be recruited into this group, their treatment will follow the standard care pathway in this observational study.
- Home HaemoDialysis (HHD) Group: Participants undergoing HHD treatment will be recruited into this group, their treatment will follow the standard care pathway in this observational study.

SUMMARY:
Individuals with kidney failure are kept alive using dialysis machines designed to remove toxic substances and excess fluid from the blood. Standard dialysis is undertaken three times a week at a dialysis unit, supported by a team of specialist dialysis nurses (so called in-centre haemodiafiltration or ICHDF). Each session lasts approximately 4 hours, during which time the fluid and toxins which have built up since the last session of treatment are removed from the blood. The rapid removal of fluid that takes place using this technique often causes unpleasant symptoms such as cramps and dizziness, as well as a "hangover", which may last several hours. It can also cause problems with the heart in the long-term.

In recent years, individuals requiring dialysis have been able to choose between standard ICHDF or having haemodialysis at home (HHD) using a convenient table top machine called NxStage System One. This device is used more frequently than in ICHDF and for shorter sessions. As a result, the amount of fluid removed during each session is less than with ICHDF. This may be beneficial to the heart, but may also make these individuals feel generally better, which may make them want to be more physically active. It may also reduce the time taken to recover from any symptoms experienced after dialysis.

Over a 12 month period, markers of heart damage (using blood tests and scans of the heart) in patients receiving frequent HHD will be studied and the results will be compared with a group of patients receiving ICHDF. The study will also compare any symptoms they may have, how fit they are, how physically active they are and how well they sleep. In addition, the investigators will assess how well fluid balance is maintained in each group and measure the changes in their remaining kidney function during this time.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HHD or ICHDF for more than 3 months and less than 36 months.
* Haemoglobin equal to or greater than100 g/L at enrolment.
* Willing and physically able to undertake the study assessments/tests
* Willing to provide blood for storage and future analysis
* Able to give informed consent

Exclusion Criteria:

* Living donor transplant or change to peritoneal dialysis planned
* Physical assessments contraindicated for the following clinical reasons

  * Acute Coronary Syndrome (ACS) within the last 3 months (chest pain, ECG changes or typical biomarker elevation).
  * Any current uncontrolled cardiac dysrhythmias causing symptoms (chest pain, palpitations, syncope or dizziness)
  * Symptomatic aortic stenosis
  * New York Heart Association grade IV Heart failure
  * Severe chronic obstructive pulmonary disease
  * Acute pulmonary embolus or pulmonary infarction in the last 3 months
  * Current acute myocarditis or pericarditis
  * Suspected or known dissecting aneurysm
  * Acute systemic infection, accompanied by fever, body aches or swollen lymph glands
* Pregnancy
* Life expectancy of less than twelve months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The start aims to recruit at the Wessex Kidney Centre, a regional renal and transplant centre based at Queen Alexandra Hospital, Portsmouth, UK (part of Portsmouth Hospitals NHS Trust). The patients involved in the study would have chosen their modality of dialysis in accordance with standard clinical practice and will not change any aspect of their treatment to meet the requirements of this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Pre- and post-dialysis levels of BNP | 12 months
  Brain Natriuretic Peptide (BNP) is one of the biomarkers of myocardial damage, it's level will be measued in EDTA anticoagulated participants' blood samples.
Pre- and post-dialysis levels of NTpro-BNP | 12 months
  N-terminal pro-brain natriuretic peptide (NTpro-BNP) is one of the biomarkers of myocardial damage, it's level will be measued in participants' serum samples.
Pre- and post-dialysis levels of TNT | 12 months
  Troponin-T (TNT) is one of the biomarkers of myocardial damage, it's level will be measued in participants' serum samples
Pre- and post-dialysis levels of Tnl | 12 months
  Troponin-L (Tnl) is one of the biomarkers of myocardial damage, it's level will be measued in participants' serum samples.
Left-ventricular mass | 12 months
  Left-ventricular mass is a well-established measure that can independently predict adverse cardiovascular events and will be determined using echocardiogram in this study
Ejection fraction | 12 months
  Visual Ejection fraction, Biplane Ejection fraction
Left ventricular global strain | 12 months
  Average GLS
Right atrial volume | 12 months
  Dertermine using echocardiogram
Integrated Back Scatter | 12 months
  Dertermine using echocardiogram

SECONDARY OUTCOMES:
Peripheral skeletal muscle oxygenation using near-infrared spectroscopy | 12 months
  Pulmonary gas exchange analyser generated data file
Maximal cardiopulmonary exercise testing (CPET) | 12 months
  Markers of physical fitness during a cycling exercise test, with concurrent measures of exercising physiological function
Breath-by-breath changes in pulmonary gas exchange and ventilation | 12 months
  Markers of physical fitness during a cycling exercise test, with concurrent measures of exercising physiological function
Objective assessment of habitual physical activity using a triaxial | 12 months
  Triaxial accelerometer generated data file consist of time went to sleep and time of waking up
Objective assessment of habitual physical activity using a triaxial accelerometer with a validated sleep diary | 12 months
  Triaxial accelerometer generated data file consist of time went to sleep and time of waking up
Blood pressure measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for blood pressure
Cardiac index measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for cardiac index
Stroke volume measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for stroke volume
Cardiac output measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for cardiac output
Total peripheral resistance measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for total peripheral resistance
Cardiac power index measued using NICOM sensor | 12 months
  Non-invasive haemodynamic measurements using NICOM sensor for cardiac power index
Concentration of pre and post dialysis Beta-2-microglobulin | 12 months
  Markers of inflammation and dialysis adequacy
Cncentration of pre-dialysis FGF-23 | 12 months
  Markers of inflammation and dialysis adequacy
Cncentration of pre-dialysis High-sensitivity CRP | 12 months
  Markers of inflammation and dialysis adequacy
Cncentration of pre-dialysis Interleukin-6 | 12 months
  Markers of inflammation and dialysis adequacy
Cncentration of pre-dialysis Interleukin-10 | 12 months
  Markers of inflammation and dialysis adequacy
Urine creatinine level | 12 months
  Residual renal function
Urine urea level | 12 months
  Residual renal function
RAPA score | 12 months
  Derivered from RAPA questionnaire
KDQoL-36 score | 12 months
  Derivered from KDQoL-36 questionnaire
FACIT-F score | 12 months
  Derivered from FACIT-F questionnaire
Recovery time | 12 months
  Patient reported recovery time after dialysis sessions and length of sleep after last dialysis session
Lean tissue mass | 12 months
  Hydration status through body composition monitoring
fat mass | 12 months
  Hydration status through body composition monitoring
Extra/intracellular water | 12 months
  Hydration status through body composition monitoring
Total body water | 12 months
  Hydration status through body composition monitoring
Saliva flow rate | 12 months
  Part of hydration status determiantion
Change in number of antihypertensive agents | Over 12 months period
  Number of antihypertensive agents
Change in erythropoietin dosage | Over 12 months period
  Erythropoietin dosage
Number of in-patient days with cause | Over 12 months period
  Date of hospital admission and date of hospital discharge
Major adverse cardiovascular events (MACE) | Over 12 months period
  Number of events considered a Major Adverse Cardiovascular Event
All-cause and cardiovascular mortality | Over 12 months period
  Number of withdrawal Information: Death of patient

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be stored anonymously once entered onto the case report form and data management database. The database will be utilised to safely and securely handle all study data and to minimise any potential risks associated with data collection. Any identifiable data, such as participant medical notes, will be kept confidential in accordance with the Caldicott Principles.